CLINICAL TRIAL: NCT05730205
Title: Effects of the Contraceptive Implant in Women With Sickle Cell Disease
Acronym: SCD CURE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 855708
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — etonogestrel; Drug Implants

STUDY DESIGN:
Intervention Model Description: Participants will be observed over two phases: 1) a 3-month phase with no hormonal contraceptive intervention and 2) a 6-month phase with the progestin implant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nexplanon (Active Comparator)
  Interventions: Drug: Nexplanon 68 MG Drug Implant
- Baseline (No Intervention)

INTERVENTIONS:
Drug: Nexplanon 68 MG Drug Implant — Progestin contraceptive device
  Arms: Nexplanon

SUMMARY:
The objective of this study is to measure the acceptability and impact of the progestin implant on frequency of vaso-occlusive crises, quality of life, and hematologic parameters in women with SCD.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is the most common inherited blood disorder in the United States, affecting 100,000 primarily Black people. The disease is characterized by chronic pain and infection, and ultimately reduces life expectancy by 20 years compared to people without SCD. Given the importance of effective contraception for women with sickle cell disease, as well as previously demonstrated therapeutic benefits of hormonal contraception, the etonogestrel implant may be an optimal method of contraception for women with SCD.

This study aims to measure the acceptability and impact of the progestin implant on frequency of vaso-occlusive crises, quality of life, and hematologic parameters in women with SCD.

This is a crossover study. Participants will be observed over two phases: 1) a 3-month phase with no hormonal contraceptive intervention and 2) a 6-month phase with the progestin implant. During the phase with no hormonal contraceptive intervention, participants must be willing to be abstinent or use a barrier method, or they must have had a permanent contraception procedure such as a tubal ligation or salpingectomy or be using the copper intrauterine device.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-45
* Diagnosis of sickle cell disease (SS or SB0)
* Report of at least 1 vaso-occlusive pain episode per month on average in the previous 6 months
* Willing to discontinue any hormonal contraception at the time of enrollment. Washout period of 1 month required for all hormonal contraception prior to enrollment in the study.
* Access to a device with text messaging capability
* Must be able to read and understand English
* Willing to comply with study procedures

Exclusion Criteria:

* SC Disease
* Use of Depo Provera in the past 6 months
* Changes to sickle cell medications in the past 3 months
* Contraindications to use of Nexplanon device as per clinical standards
* Currently pregnant or pregnant within the last month or seeking to become pregnant
* Currently breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of vaso-occlusive crises | 9 months
  Self-reported pain crises, discrete pain episodes will be separated by at least 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine University City, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No